CLINICAL TRIAL: NCT03634397
Title: Predicting Ipsilesional Motor Deficits in Stroke With Dynamic Dominance Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert L. Sainburg (Other)
Collaborators: University of Southern California (Other); Penn State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Robert L. Sainburg, Professor of Kinesiology and Neurology, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008385; R01HD059783-06A1 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2018-08-16 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups. One group (treatment group) receives remediation therapy of the less impaired arm while the control group receives paretic arm therapy.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will assess all participants and be unaware of the participants' group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Less-Impaired Arm Training (Experimental): Intervention condition includes therapy of the less-impaired (ipsilesional) arm.
  Interventions: Behavioral: Less-Impaired Arm Training
- Contralesional Arm Comparison (Sham Comparator): Comparison control condition includes therapy of the paretic (contralesional) arm.
  Interventions: Behavioral: Contralesional Arm Comparison

INTERVENTIONS:
Behavioral: Less-Impaired Arm Training — Participants receive virtual reality and manipulation training in their less impaired arm.
  Arms: Less-Impaired Arm Training
Behavioral: Contralesional Arm Comparison — Participants receive therapy in their paretic arm, based on the best-practices framework for arm recovery post stroke.
  Other Names: sham condition
  Arms: Contralesional Arm Comparison

SUMMARY:
This study will test the hypothesis that the combination of low-moderate to severe motor deficits in the paretic arm and persistent motor deficits in the less-impaired arm limits functional independence in chronic stroke survivors. We, therefore, predict that intense remediation, focused on improving the speed, coordination, and accuracy of the less-impaired arm should improve functional independence.

DETAILED DESCRIPTION:
We previously characterized hemisphere-specific motor control deficits in the non-paretic arm of unilaterally lesioned stroke survivors. Our preliminary data indicate these deficits are substantial and functionally limiting in patients with severe paresis. We have specifically designed an intervention to remediate the hemisphere-specific deficits in the less-impaired arm, using a virtual-reality platform, and then follow this training with manipulation training of a variety of real objects, designed to facilitate generalization and transfer to functional behaviors encountered in the natural environment. We propose a 2-site, two-group randomized intervention with a treatment group, which will receive unilateral training of the less-impaired arm, through our Virtual Reality and Manipulation Training (VRMT) protocol. This intervention protocol is grounded in the premise that targeted remediation of fundamental control deficits exhibited by the less-impaired arm will generalize and transfer beyond practiced tasks to performance of activities of daily living (ADL). This approach contrasts with the more pragmatic approach of task-specific training of essential ADL's, which is limited in scope, more cumbersome, and ignores known fundamental motor control deficits. Our control group will receive conventional intervention, guided by recently released practice guidelines for upper limb intervention in adult stroke. The impact of the proposed research is that we address persistent functional performance deficits in chronic stroke patients with severe paresis, who's less-impaired arm impairments are generally ignored in most current rehabilitation protocols. Our first aim addresses the overall effectiveness of this intervention, relative to our control group: To determine whether non-paretic arm VRMT in chronic stroke survivors with severe paresis will produce durable improvements in less-impaired arm motor performance that will generalize to improve functional activities and functional independence to a greater extent than conventional therapy focused on the paretic arm. Our second aim focuses on the mechanistic basis of potential training-related improvements in motor performance: To determine whether intervention-induced improvements in less-impaired arm performance are associated with improvements in hemisphere-specific reaching kinematics. Finally, our third aim monitors for potential negative effects of our experimental intervention on paretic arm impairment.

ELIGIBILITY:
Inclusion Criteria:

1. neuroradiological confirmation of unilateral brain damage with residual contralesional upper-extremity weakness
2. deficits in ipsilesional arm performance assessed by the JTHFT
3. 6+ months post stroke
4. Demonstrates cognitive abilities

Exclusion Criteria:

a history of:

1. neurological disease other than stroke (e.g., head trauma)
2. a major psychiatric diagnosis (e.g., schizophrenia, major affective disorder),
3. hospital admission for substance abuse
4. peripheral disorders affecting sensation or movement of the upper extremities, including pain or arthritis
5. currently taking prescription drugs with known sedative properties that are interfering with sensory-motor function
6. significant joint pain that is activity limiting
7. bilateral stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Sainburg, Phd, OTR, Principal Investigator — Penn State University; Carolee J Winstein, PhD,PT, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Penn State College of Medicine, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data (functional outcome measures) generated by the project will be shared through ScholarSphere (https://scholarsphere.psu.edu/), the repository service that both the University Libraries and Information Technology Services administer at Penn State. Researchers will be able to access the data via ScholarSphere, which ensures persistent access to deposited content. The data will be discoverable via Google and other major search engines, as well as by request to Dr. Sainburg or Dr. Winstein.
Time Frame: Within one year of study completion, available for a minimum of one year.
Access Criteria: The web address is open to the public.
URL: https://scholarsphere.psu.edu/

REFERENCES:
- [Derived] Maenza C, Winstein CJ, Murphy TE, Kitchen NM, Tanaka J, Yuk J, Varghese R, Sainburg RL. Targeted Remediation of the Ipsilesional Arm in Chronic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2026 Feb 2:e255496. doi: 10.1001/jamaneurol.2025.5496. Online ahead of print. PMID 41627841
- [Derived] Maenza C, Sainburg RL, Varghese R, Dexheimer B, Demers M, Bishop L, Jayasinghe SAL, Wagstaff DA, Winstein C; IPSI Investigative Team. Ipsilesional arm training in severe stroke to improve functional independence (IPSI): phase II protocol. BMC Neurol. 2022 Apr 12;22(1):141. doi: 10.1186/s12883-022-02643-z. PMID 35413856

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipsilesional Arm Training (Experimental Condition): Intervention condition includes therapy of the less-impaired (ipsilesional) arm.
  Ipsilesional (Less-Impaired) Arm Training: Participants receive virtual reality and manipulation training in their less impaired arm.
- Contralesional Arm (Comparison Condition): Comparison control condition includes therapy of the paretic (contralesional) arm.
  Contralesional Arm Comparison: Participants receive therapy in their paretic arm, based on the best-practices framework for arm recovery post stroke, for the same duration as the experimental ipsilesional arm training condition.
Period: Overall Study
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Started | 29 | 29
Completed | 25 | 28
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ipsilesional Arm Training (Experimental Condition): Intervention condition includes therapy of the less-impaired ipsilesional arm.
  Ipsilesional Arm Training: Participants receive virtual reality and manipulation training in their less impaired arm.
- Contralesional Arm (Comparison Condition): Comparison control condition includes therapy of the paretic (contralesional) arm.
  Contralesional Arm Comparison: Participants receive therapy in their paretic arm, based on the best-practices framework for arm recovery post stroke.
- Total: Total of all reporting groups
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 58 [30 to 74] | 59 [40 to 81] | 59 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 23 | 23 | 46
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
Jebsen-Taylor Hand Function Test [Count of Participants; unit: Participants] | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Jebsen-Taylor Hand Function Test (JTHFT) Times From Baseline 2 to Post Test 1
Description: Measure of unimanual arm performance in a wide range of hand functions required for activities of daily living. The test includes 7 timed (seconds) activities (possible 0-120 seconds each); the analysis excludes the writing component, therefore it includes 6 of the 7 original JTHFT components. Faster performance yields lower scores (time).
  There were 2 baseline tests (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score as the starting value and do not include the first baseline scores.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: 5 participants were randomized, but did not complete intervention due to Covid epidemic, and thus did not have JTHFT at post test 1.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 25 | 28
seconds | 5.07 (.93) | -.11 (1.37)
Statistical Analysis 1: Comparison: Ipsilesional Arm Training (Experimental Condition) vs Contralesional Arm (Comparison Condition); Test type: Other; p < .05, Regression, Linear — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; Mean Difference (Final Values) = 5.73, 95% CI 2-sided [2.31 to 9.14] — The delta values of the outcome from baseline 2 to post-treatment 1 were directly modeled using linear regression with adjustment for age, female sex, and the hemisphere affected by the stroke

2. Primary Outcome: Change in Abilhand Scores From Baseline 2 (Prior to Treatment) to Post Test 1
Description: Participant reported outcome of difficulty of upper extremity based activities. Scores are transformed to logit scores. The items ranged on the interval scale from -2.18 to 1.72 log-odds units, called 'logits', with higher logit values indicating more difficult activities. Deltas of logits from baseline 2 to post test 1 are reported. There were two baseline assessments (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score (when participants were randomized) as the starting value and do not include the first baseline scores. Results do not include covariates.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: All participants with baseline 2 and post test 1 data were included in analysis. Scores are transformed to logit scores. The items ranged on the interval scale from -2.18 to 1.72 log-odds units, called 'logits', with higher logit values indicating more difficult activities. Deltas of logits from baseline 2 to post test 1 are reported.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 25 | 28
score on a scale | -2.08 (1.43) | -.57 (1.18)

3. Primary Outcome: Change of Score on Barthel Index From Baseline 2 (Prior to Training) to Post Test 1
Description: Measure of functional independence in self care activities scored from 0-100 with higher scores indicating more functional independence. There were two baseline assessments (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score (when participants were randomized) as the starting value and do not include the first baseline scores.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: Only participants with baseline 2 and post test 1 are included in analysis. Delta values from baseline 2 to post test 1 are reported and adjusted for age, sex, and hemisphere of lesion.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 25 | 28
score on a scale | -1.2 (1.83) | -1.79 (1.24)
Statistical Analysis 1: Comparison: Ipsilesional Arm Training (Experimental Condition) vs Contralesional Arm (Comparison Condition); Test type: Other — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; p < .05, Regression, Linear — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; Mean Difference (Final Values) = .83, 95% CI 2-sided [-2.58 to 4.24]

4. Primary Outcome: Change in Upper-Extremity Fugl-Meyer Assessment (FM) Score From Baseline 2 (Prior to Training) to Post Test 1
Description: Upper-Extremity Measure of paretic arm impairment out of 66 possible points with higher scores indicating more movement, and 0 indicating no functional movement in the arm. There were two baseline assessments (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score (when participants were randomized) as the starting value and do not include the first baseline scores.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: Only participants with data at baseline 2 and post test 1 are included in analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 25 | 28
score on a scale | -.68 (.8) | -1.61 (.93)
Statistical Analysis 1: Comparison: Ipsilesional Arm Training (Experimental Condition) vs Contralesional Arm (Comparison Condition); Test type: Other — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; p < .05, Regression, Linear — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke; Median Difference (Final Values) = 1.12, 95% CI 2-sided [-2.29 to 4.53] — P-values include adjustment for age, female sex, and hemisphere of brain affected by stroke

5. Secondary Outcome: Change From Baseline 2 (Prior to Training) to Post Test 1on Functional Independence Measure (FIM) -Self Care Components
Description: Each item on the FIM is scored on a 7-point Likert scale, and the score indicates the amount of assistance required to perform each item (1 = total assistance in all areas, 7 = total independence in all areas). Analysis includes 6 sub-components of the FIM, which are the self care components (Eating, Grooming, Bathing, Dressing upper body, Dressing lower body, and toileting) (possible 42 points). Higher scores indicate more independence.
  There were two baseline tests (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score as the starting value and do not include the first baseline scores.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: All participants with baseline 2 and post test 1 data were analyzed (N=53). 5 randomized participants were excluded from analysis because they did not have baseline 2 and post test 1 measures due to Covid disruption.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 25 | 28
score on a scale | -1.44 (.75) | -.46 (.81)

6. Secondary Outcome: Change From Baseline 2 (Prior to Training) to Post Test 1 on Contralesional Work Space Area (Kinematics)
Description: Workspace area is a kinematic measure of active range of motion, which we measured on the paretic (contralesional) arm. This was calculated by computing the area of the ellipse (measured in centimeters) formed by the major and minor axis of the contralesional arm trajectory on each trial. The major axis was defined as the largest distance between any two points in the handpath, while the minor axis was defined as the largest distance, perpendicular to the major axis. Values were averaged within subjects over all trials for each evaluation (i.e. BL2 and PT1), then group and evaluation averages and standard deviations were calculated from these values.
  There were two baseline tests (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score as the starting value and do not include the first baseline scores. These values do not include covariates.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: Participants were excluded from this analysis if they could not complete the kinematics for any reason (i.e.: Covid, a pacemaker, not fitting in the kinematic setup), or did not complete both baseline and post test 1 kinematic assessments.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 21 | 26
centimeters | 0.512 (2.1217) | 0.340 (1.6714)

7. Secondary Outcome: Change in Kinematics- Positional Variability at Maximum Velocity From Baseline 2 (Prior to Training) to Post Test 1
Description: Positional variability is a measure of kinematic variability in reaching movement. This was measured at the participants max reaching velocity and their end position. This was calculated by taking the distance (cm) from the fingertips location at peak velocity/end position on a given trial from its mean location at peak velocity/end position across all trials, for each target. Values were averaged within subjects over all trials for each evaluation (i.e. BL2 and PT1), then group and evaluation averages and standard deviations were calculated from these values.
  There were two baseline tests (3 weeks apart) to show unchanged performance in assessments prior to training. Training included 15 sessions over the course of up to 7 weeks. Results reported used the second baseline score as the starting value and do not include the first baseline scores or covariates.
Time Frame: Baseline 2 to Post Test 1 (up to 2 weeks post last treatment session)
Population: Participants were excluded if they could not complete the kinematic portion of the study due to Covid, or a pacemaker, or not fitting in the kinematic setup, or if they didn't complete both baseline and post test 1 assessments.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
Number analyzed (Participants) | 21 | 26
Centimeters
  Maximum Velocity | 0.0930727 (0.4369149) | -0.0225708 (0.4979299)
  End Position | 0.2811583 (0.5066384) | -0.1156399 (1.1076122)

ADVERSE EVENTS:
Time Frame: Over the course of the study, up to 12 months following study enrollment.
Arm/Group | Ipsilesional Arm Training (Experimental Condition) | Contralesional Arm (Comparison Condition)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/29
Other Adverse Events (participants affected / at risk) | 2/29 | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipsilesional Arm Training (Experimental Condition) (N=29) | Contralesional Arm (Comparison Condition) (N=29)
Pain resulting in hospitalization (General disorders) | 1 (1) | 0 (0)
Fall with knee injury (General disorders) | 0 (0) | 1 (1) — Resulted in hospitalization, unrelated to the study
Hit head (outside of the intervention period) (General disorders) | 1 (1) | 0 (0) — Event occurred outside of the study, but prior to completing a post test.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipsilesional Arm Training (Experimental Condition) (N=29) | Contralesional Arm (Comparison Condition) (N=29)
back pain (General disorders) | 0 (0) | 1 (1)
kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
chronic depressive symptoms (Psychiatric disorders) | 0 (0) | 2 (2)
fall with no fracture (General disorders) | 0 (0) | 1 (1)
benign growth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was ongoing during the start of the Covid epidemic and the laboratory was shut down for an extended period of time resulted in lower than expected number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03634397/Prot_SAP_000.pdf